CLINICAL TRIAL: NCT03598517
Title: Intensity-modulated Hyperfractionated Radiotherapy Boost to Residual Metabolic Disease Following Standard Chemoradiotherapy for Locally Advanced Non-small Cell Lung Cancer
Brief Title: High Dose Radiation Therapy With Concurrent Chemotherapy in Locally Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chen tingfeng, director, department of radiation, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGH201816
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- high dose chemoradiotherapy (Experimental): all eligible patients receive image-guided intensity-modulated radiotherapy 60 Gy in 30 fractions over 6 weeks and concurrent weekly paclitaxel and cisplatin，followed by hyperfractionated intensity-modulated radiotherapy boost to residual metabolic disease concurrent with the same chemotherapy regimen, followed by adjuvant chemotherapy 6 weeks after completion of radiation therapy.
  Interventions: Radiation: high dose chemoradiotherapy

INTERVENTIONS:
Radiation: high dose chemoradiotherapy — Radiation therapy: 60 Gy at 2 Gy/Fx/d over 6 weeks, immediately followed by 28.8 Gy in 24 fractions of 1.2 Gy, twice per day,on weeks 6-8 to a total dose of 88.8 Gy.
  concurrent chemotherapy: weekly carboplatin area under the curve (AUC) 2 and paclitaxel 45 mg/m2 over the duration (8 weeks) of radiation therapy.
  Adjuvant chemotherapy is planned 6 weeks after high dose chemoradiation.

SUMMARY:
To assess the efficacy and feasibility of high-dose intensity-modulated radiotherapy with concurrent weekly paclitaxel and cisplatin for patients with locoregionally advanced non-small lung cancer.

DETAILED DESCRIPTION:
Local failure remains high in patients with locoregionally advanced non-small lung cancer. Given that a biological equivalent dose (BED)more than 100 Gy yields approximately a local control rate of 90% in early-stage non-small lung cancer, this BED or ever higher is logically required to control local disease for locally advanced non-small lung cancer. However, dose escalation is limited by radiation-related toxicity. Use of hyperfractionated radiation Therapy boost to residual metabolic disease as defined by positron emission tomography and computed tomography (PET/CT) immediately after standard chemoradiotherapy (SCRT) using image-guided (IG) IMRT could potentially improve local control and perhaps survival

ELIGIBILITY:
Inclusion Criteria:

* Patients must have FDG-avid and histologically or cytologically proven non-small cell lung cancer.
* Age 1 8-75.
* Eastern Cooperative Oncology Group （ECOG） performance status 0 to 2.
* Stage III ( American Joint Committee on Cancer AJCC, 7th ed.).
* No prior radiation to the thorax that would overlap with the current treatment field.
* Adequate bone marrow, renal and hepatic functions as assessed by the following: Hemoglobin >/= 10.0 g/dl, Platelet count >/= 1 00,000/ mm^3,absolute granulocyte count (AGC) ≥2 × 10^9 cells/L,bilirubin and Aspartate transaminase ≤1.5 ×upper limit of normal (ULN), Creatinine </ =1 .5 times ULN.
* A signed informed consent must be obtained prior to therapy.
* Induction chemotherapy is allowed.
* Life expectancy more than 3 months

Exclusion Criteria:

* Patients with any component of small cell lung carcinoma are excluded from this study.
* Patients with evidence of a malignant pleural or pericardial effusion are excluded.
* Prior radiotherapy that would overlap the radiation fields.
* Uncontrolled concurrent illness including, but not limited to: Chronic Obstructive Pulmonary Disease(COPD) exacerbation or other respiratory illness, serious uncontrolled infection, symptomatic congestive heart failure (CHF),unstable angina pectoris, uncontrolled hypertension,or psychiatric illness/social situations that would limit compliance with the study requirements.
* Known hypersensitivity to paclitaxel.
* Any other condition or circumstance that would, in the opinion of the Investigator, make the patient unsuitable for participation in the study.
* Conditions precluding medical follow-up and protocol compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
overall survival rate | 2 year
  survival time was measured from the date of study enrollment to the date of death or last follow-up

SECONDARY OUTCOMES:
toxicities | 2 year
  Acute toxicities were graded according to the National Cancer Institute-Common Toxicity Criteria (NCI-CTC) version 4.

CONTACTS AND LOCATIONS:
Overall Officials: Tingfeng Chen, MD, Study Director — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Genernal Hospital, Shanghai, Shanghai Municipality, China